CLINICAL TRIAL: NCT00640458
Title: A Double Blind, Placebo Controlled 2-way Cross-over Study to Assess the Clitoral Engorgement Response as Measured by Non-contrast Magnetic Resonance Imaging (MRI) in Women With Female Sexual Arousal Disorder (FSAD) When Administered a Single Dose of Sildenafil (100mg) Followed by Audio/Visual Sexual Stimulation
Brief Title: Study to Investigate Effect of Sildenafil on Clitoral Engorgement as Measured by Magnetic Resonance Imaging (MRI) in Pre-menopausal Women With Female Sexual Arousal Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: A1481174
Record Dates: First submitted 2008-03-17; First posted 2008-03-21 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Female Sexual Arousal Disorder
MeSH Terms: interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Study Period 1 or 2
  Interventions: Drug: Placebo
- Experimental (Experimental): Study Period 1 or 2
  Interventions: Drug: Sildenafil 100 mg

INTERVENTIONS:
Drug: Sildenafil 100 mg
  Arms: Experimental
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the effect of 100 mg sildenafil on clitoral engorgement in pre-menopausal women, as well as examining the safety and toleration of the drug.

ELIGIBILITY:
Inclusion Criteria:

* Pre-menopausal women aged 18-45 with a primary diagnosis of Female Sexual Arousal Disorder for at least 6 months prior to entering the study. The FSAD could have been associated with female orgasmic disorder (FOD) and/or superficial or introital dyspareunia.

Exclusion Criteria:

* Subjects with hypoactive sexual desire disorder.
* Subjects not using an acceptable mean of contraception for the duration of the study.
* Subjects who were prescribed and/or taking medication which were contraindicated or cautioned with concomitant intake of sildenafil.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2004-04; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
To determine the % of subjects who respond within 30 minutes of dosing by achieving an increase in clitoral engorgement >50% from baseline measured by MRI following audio/visual sexual stimulation in females with FSAD. | Up to 30 minutes post-dose

SECONDARY OUTCOMES:
To determine the % of subjects who respond to sildenafil 100mg by achieving an increase in clitoral engorgement >50% from baseline within 40, 50 and 60 minutes of dosing respectively. | Up to 60 minutes post-dose
To assess safety and toleration of sildenafil 100mg by adverse event monitoring, laboratory safety testing and physical examination findings. | 30 days post-dose
Assess plasma levels of sildenafil and metabolite | Day of dosing

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- Pfizer Investigational Site, Seattle, Washington, United States
- Pfizer Investigational Site, Nedlands, Western Australia, Australia

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1481174&StudyName=Study%20to%20investigate%20effect%20of%20sildenafil%20on%20clitoral%20engorgement%20as%20measured%20by%20magnetic%20resonance%20imaging%20%28MRI%29%20in%20pre-menopausal%20wo